CLINICAL TRIAL: NCT03946943
Title: A Single-arm, Single-center Prospective Study of Anlotinib Hydrochloride and Toripalimab in Subjects With Unresectable or Metastatic Undifferentiated Pleomorphic Sarcoma Patients
Brief Title: Study of Anlotinib Hydrochloride and Toripalimab in Subjects With Unresectable or Metastatic Undifferentiated Pleomorphic Sarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Di Wu (Other)
Responsible Party: Sponsor-Investigator, Di Wu, chief, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FHJLU-003
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Soft Tissue Sarcomas; Undifferentiated Pleomorphic Sarcoma
Keywords: TKI; PD-1 inhibitor; Anlotinib
MeSH Terms: conditions — Sarcoma; Histiocytoma, Malignant Fibrous | interventions — anlotinib; toripalimab; Blood Specimen Collection; Phlebotomy; Biopsy, Needle

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anlotinib + Toripalimab (Experimental): Concurrent anlotinib and Toripalimab therapy, with Blood Draw and Tumor Specimen Collection for correlative studies
  Interventions: Drug: Anlotinib; Drug: Toripalimab; Procedure: Blood Draw; Procedure: Tumor Specimen Collection

INTERVENTIONS:
Drug: Anlotinib — Once a day dosing of anlotinib alone for the first 7 days, Anlotinib ( 12mg, QD, PO, d1-14, 21 days per cycle), take once when limosis in the morning. If patients cannot suffer from AEs, they can get declined dosage.
Drug: Toripalimab — Toripalimab 240mg shall be administered via intravenous (IV) infusion, once every 21 days, on day 8 and day 29 of the first cycle, and days 1 and 22 of the following cycles.
Procedure: Blood Draw — Peripheral blood draws for correlative studies characterizing T-cells in peripheral blood will be performed at three timepoints: 1) pre-treatment, 2) on-treatment on cycle 3 day 1, and 3) off-study.
  Other Names: Phlebotomy
Procedure: Tumor Specimen Collection — Tumor specimen collection via core needle biopsy for correlative studies characterizing T-cells in tumor tissue will occur at three timepoints: 1) pre-treatment, 2) on-treatment on cycle 3 day 1, and 3) off-study.
  Other Names: Core-Needle Biopsy

SUMMARY:
The investigators hypothesize that combination anlotinib with toripalimab will improve progression-free survival relative to historical controls in patients with Unresectable or Metastatic Undifferentiated Pleomorphic Sarcoma.

DETAILED DESCRIPTION:
This is a single-institution, open-label, single-arm Phase II study to determine the efficacy and safety of anlotinib in combination with Toripalimab compared with historical controls as first-line treatment in patients with Unresectable or Metastatic Undifferentiated Pleomorphic Sarcoma.

Since the primary endpoint is survival outcome, progression-free survival (PFS) sample size calculation is based on a single-arm survival design. The investigators will employ early stopping rules for lack of efficacy, based on previously reported historical controls progression-free rate at 3 months was 57% in MFH and This study predicts that as the First-Line treatment of Undifferentiated Pleomorphic Sarcoma, progression-free rate at 3 months is expected to reach more than 80%.

Patients will be treated with once a day dosing of anlotinib alone for the first 7 days, followed by concurrent anlotinib administered once a day at 12mg orally (PO), plus intravenous administration of toripalimab every 21 days. Patients will be assessed every six weeks for toxicity. After the first five patients are enrolled, the investigators will assess safety of the combination. If 2 or fewer patients exhibit dose-limiting toxicity (DLT), the investigators will then proceed with intrapatient titration of anlotinib dosing at each cycle based on the presence or absence of predefined toxicities.

Correlative studies characterizing T-cells in tumor tissue and in peripheral blood will be performed at three timepoints: 1. pre-treatment, 2. on-treatment on cycle 3 day 1, and 3. off-study. Additional exploratory imaging investigations, and assessment of circulating tumor cells are included for all patients.

Trial therapy will last until withdrawal of consent, disease progression and/or unacceptable toxicity, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed Undifferentiated Pleomorphic Sarcoma with pathology review required for any outside samples.

   Only patients with untreated and rejected first-line standard chemotherapy with high-grade Undifferentiated Pleomorphic Sarcoma can be enrolled
2. Any other histology or standard of care therapy not specifically addressed will be reviewed by the principal investigator and pathologist for final determination of eligibility.
3. Measurable disease as defined by RECIST v1.1
4. Radiographic progression as defined by RECIST v1.1, based on comparison between two radiographic studies no greater than 3 months apart. or Inability to undergo complete resection of the disease by surgery.
5. Adequate organ function as defined:

   Hematological
   1. Absolute neutrophil count (ANC) ≥1,000 / microliter (mcL)
   2. Platelets ≥75,000 / mcL
   3. Hemoglobin ≥8 g/dL without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment)

   Renal

   Serum creatinine ≤1.5 X upper limit of normal (ULN) OR Measured or calculated creatinine clearance ≥ 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN. (GFR can also be used in place of creatinine or CrCl). Creatinine clearance should be calculated per institutional standard.

   Hepatic
   1. Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN.
   2. Aspartate Aminotransferase (AST/SGOT) and Alanine Transaminase (ALT/SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases.
   3. Albumin >2.5 mg/dL

   Coagulation
   1. International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
   2. Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
6. Age ≥ 16 years.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. Expected Survival Time: Over 3 months;
9. Patients must consent and be willing to undergo three core needle biopsies at baseline, prior to starting Cycle 3, and at off-study. At least one tumor site must be amenable to biopsy in the judgment of the interventional radiologist.
10. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
11. Females of child bearing potential that are sexually active must agree to either practice 2 medically accepted highly effective methods of contraception at the same time or abstain from heterosexual intercourse from the time of signing the informed consent through 120 days after the last dose of study drug. See Appendix G for protocol-approved highly effective methods of contraceptive combinations. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.

    1. Negative test for pregnancy is required of females of child-bearing potential; A female of child bearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1. has not undergone a hysterectomy or bilateral oophorectomy; or 2. has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months or 730 days).
    2. Conception while on treatment must be avoided
12. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy. Prior history of vasectomy does NOT replace requirement for contraceptive use.
13. Suitable venous access to allow for all study related blood sampling
14. Ability to understand and willingness to sign a written informed consent document.
15. For minors that are 16 to 18 years of age, assent and parental (or legally acceptable representative) written informed consent must be obtained.

Exclusion Criteria:

1. Prior therapy with anlotinib. Patients who have received prior tyrosine kinase inhibitor (TKI) therapy including imatinib, sunitinib, pazopanib, or similar. Patients who have received immunotherapy including Programmed death 1 (PD-1)/Programmed death-ligand 1 (PD-L1) and CTLA-4.
2. Hypersensitivity to anlotinib, pembrolizumab or any of its excipients.
3. Patients may not be receiving any other investigational agents (within 4 weeks prior to Cycle 1, day 1).
4. If subject received palliative surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
5. Additional known malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, or squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cervical cancer.
6. Patients with end-organ dysfunction as defined in inclusion criterion (i.e. #6 above).
7. Patients with bone-only lesions.
8. Patients with underlying immune deficiency, chronic infections including HIV, hepatitis, or tuberculosis (TB) or autoimmune disease.
9. Any major unhealed wound, ulcer, or fracture occurred in a patient who had undergone major surgery or trauma within 4 weeks and/or had any bleeding or bleeding episodes which the degree is bigger than CTCAE 3 grade within 4 weeks prior to enrollment.
10. Arteriovenous thrombosis events occurred within 6 months. Such as cerebrovascular accidents (including transient ischemic attacks), deep vein thrombosis and pulmonary embolism
11. History of steroid-related (non-infectious) pneumonia or current pneumonia.
12. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis or leptomeningeal disease. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
13. Concomitant (or receipt of) treatment with medications that may affect the metabolism of pembrolizumab and/or axitinib within 7 days prior to Cycle 1, day 1 of anlotinib.
14. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
15. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
16. Any uncontrolled, intercurrent illness including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia
17. rolonged corrected QT (QTc) interval on Screening EKG >475 ms. Ejection Fraction <40% by 2D echocardiogram (ECHO) at Screening.
18. Any serious medical or psychiatric illness/condition including substance use disorders likely in the judgment of the Investigator(s) to interfere or limit compliance with study requirements/treatment.
19. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-07-19 (Estimated); Primary Completion 2022-07-19 (Estimated); Study Completion 2023-07-19 (Estimated)

PRIMARY OUTCOMES:
Rate of Participants Achieving 3-Month Progression-Free Survival (PFS) | 3 Months after start of protocol therapy
  Rate of participants who are progression-free at 3 months after the start of protocol therapy, using Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 criteria. Progression-free survival (PFS) is defined as the time from treatment initiation until documented disease progression or death (by any cause, in the absence of progression).

SECONDARY OUTCOMES:
Rate of Participants Achieving 6-Month and 12-Month Progression-Free Survival (PFS) | 6 Months and 12 Months after start of protocol therapy
  Rate of participants who are progression-free at 6 months and 12-Month after the start of protocol therapy, using Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 criteria.
Rate of Participants Achieving Objective Response (ORR) | 3, 6, and 12 Months after start of protocol therapy
  Rate of participants achieving complete response (CR) or partial response (PR) at 3, 6 and 12 months after the start of protocol therapy, according to RECIST version 1.1 criteria.
Rate of Participants Achieving Clinical Benefit (CBR) | 3, 6, and 12 Months after the start of protocol therapy
  Rate of participants achieving complete response (CR), partial response (PR) or stable disease (SD) at 3, 6 and 12 months after the start of protocol therapy, according to RECIST version 1.1 criteria.
Duration of Response（DOR） | up to two year
  Defined as the time between the first assessment of a tumor as PR or CR and the first assessment as PD or any cause of death，according to RECIST version 1.1 criteria.
Time to initial Response（TTR） | up to two year
  Defined as the time between participant enrollment to the first assessment of a tumor as PR or CR，according to RECIST version 1.1 criteria.
Overall Survival (OS) | Through Study Completion, an Average of 12 months
  Defined as the time between participant enrollment to death or date of censoring.
Safety and Toxicity Profile: Rate of Toxicity in Study Participants | Up to 30 days after the end of protocol therapy
  Rate of dose-limiting toxicities (DLTs) and/or grade 3 or 4 serious adverse events (SAEs) in study participants up to 30 days after the end of protocol therapy. Toxicity will be assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

OTHER OUTCOMES:
Change in quantity of CD3+ T-cells in Peripheral Blood and Tumor Tissue | Baseline, cycle 3, and off-study, an Average of 12 months
  The quantity of CD3+ T-cells in peripheral blood and in tumor biopsies at each timepoint (baseline, cycle 3, and off-study).
Expression Category of T-cell subsets in Tumor Tissue | Baseline, cycle 3, and off-study, an Average of 12 months
  The expression category in tumor tissue (none (0%), low (<5%), intermediate (5-50%), or high (>50%) of PD-1, PD-L1, PD-L2, CTLA-4, TIM-3, LAG-3 at each timepoint (baseline, cycle 3, and off-study).
Absolute Change in T-cell Marker Levels in Peripheral Blood and Tumor Tissue | Baseline, Cycle 3, Progression, an Average of 12 months
  The following T cell subsets will be studied in peripheral blood and tumor tissue: (CD4, CD8, T-reg, CTLA4, TIM3, LAG3, memory, naïve, PD-1, Ki67). For each marker, the absolute change in the marker(s) value will be calculated:
  1. Cycle 3 marker value minus Baseline marker value
  2. Progression marker value minus Cycle 3 marker value
  3. Progression marker value minus Baseline marker value
Description of the Relationship between tumor response according to RECIST 1.1 and tumor response according to alternative radiologic methods | Baseline, Cycle 3, off-study, an Average of 12 months
  Utilizing each of the alternative (non-RECIST) radiological criteria the investigators will categorize clinical benefit status (CR/PR/SD vs PD). CT and/or MRI with dynamic contrast enhanced sequences will be collected throughout the study at every disease evaluation and analyzed using Choi criteria, MRI volumetrics, and immune-related response criteria. PET/CT will be obtained at baseline, Cycle 3, and off-study and tumor response determined by Positron Emission Tomography (PET) Response Criteria in Solid Tumors (PERCIST 1.0).
Change in Quantity of Circulating Tumor Cells (CTCs) in Peripheral Blood | Baseline, Cycle 3, and Off-study, an Average of 12 months
  The quantity of circulating tumor cells (CTCs) in peripheral blood will be measured at three timepoints: baseline, cycle 3, and off-study.

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China

REFERENCES:
- [Background] Van Glabbeke M, Verweij J, Judson I, Nielsen OS; EORTC Soft Tissue and Bone Sarcoma Group. Progression-free rate as the principal end-point for phase II trials in soft-tissue sarcomas. Eur J Cancer. 2002 Mar;38(4):543-9. doi: 10.1016/s0959-8049(01)00398-7. PMID 11872347